CLINICAL TRIAL: NCT05971667
Title: "Effect of Tadalafil, Sildenafil and Pentoxyfylline on Endometrial Thickness and Frozen Embryo Transfer Outcomes
Brief Title: Effect of Tadalafil, Sildenafil and Pentoxyfylline on Frozen Embryo Transfer Outcomes
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sara Abdallah Mohamed Salem, Lecturer of Gynecology and obstetrics Faculty of medicine Beni-Suef University, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tadalafil IVF
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: IVF
Keywords: Tadalafil; Sildenafil; pentoxyfylline; frozen embryo transfer
MeSH Terms: interventions — Tadalafil; Sildenafil Citrate; Pentoxifylline

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- tadalafil (Experimental): tadalafil 10 mg one tablet daily
  Interventions: Drug: tadalafil
- pentoxifylline (Experimental): pentoxyfilline 400 mg two tabs daily
  Interventions: Drug: pentoxifylline
- sildenafil (Experimental): sildenafil 20 mg two tablets
  Interventions: Drug: Sildenafil
- control group. (No Intervention): no intervention is given

INTERVENTIONS:
Drug: tadalafil — tadalafil 10 mg one tablet daily
  Other Names: cialong
  Arms: tadalafil
Drug: Sildenafil — sildenafil 20 mg two tablets daily
  Other Names: Respatio
  Arms: sildenafil
Drug: pentoxifylline — pentoxifylline 400 mg two tabs daily
  Other Names: trental
  Arms: pentoxifylline

SUMMARY:
The aim of this study is to investigate the Effect of different vasodilators as Tadalafil, Sildenafil and pentoxyfylline in In vitro Fertilization. In addition, the thickness of endometrium and pregnancies rates of these women will also be examined. All adverse effects of all drugs will be estimated

DETAILED DESCRIPTION:
A prospective randomized clinical study will be conducted in the IVF clinic of the gynecology department of Beni Suef University Hospital, Beni-Suef, Egypt. The study will These patients will be randomized into four groups.

The participants will take drugs starting from the end of menstruation cycle till endometrium reach optimal and then will start progesterone 800 mg daily.

ELIGIBILITY:
Inclusion Criteria:

* women having thawed embryos

Exclusion Criteria:

* hypotension
* cardiovascular, hepatic, and renal diseases;
* uncontrolled diabetes mellitus;
* ovarian cysts;
* hyperprolactinemia;
* abnormal thyroid functions;
* uterine fibroids;
* patients taking nitrates;
* endometriosis and adenomyosis

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-07-30 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
endometrial thickness | within 16 day of menstruation
  measured by transvaginal ultrasound

SECONDARY OUTCOMES:
pregnancy rate | 1 month
  number of cases positive serum pregnancy test

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-suef university Hospital, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided